CLINICAL TRIAL: NCT01878851
Title: Characterization of Blood Drawn From the Pulp of Primary Molar Undergoing Pulpotomy or Pulpectomy.
Status: Withdrawn | Type: Observational
Why Stopped: New data was published in the literature
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Moti Moskovitz, Senior Clinical Lecturer, Hadassah Medical Organization
Other Study IDs: Moti-Kot-HMO-CTIL
Record Dates: First submitted 2013-06-13; First posted 2013-06-17 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Inflammatory Markers; Pulpotomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pulpotomy

SUMMARY:
Following medical history and clinical examination the children which are scheduled for treatment with suspected pulpary involved primary teeth will be selected. During the regular treatment if a pulp of primary teeth is opened and before the regular pulpotomy procedure is performed the blood that is flowing out of the pulp will be collected and stored until analyzed for the present of inflammatory markers. Clinical and radiographic evaluation will be obtained in follow up appointments if the child will remain in regular treatments in our clinic.

ELIGIBILITY:
Inclusion Criteria:

- Pulpal involved primary teeth with a vital pulp of which a certain amount of blood can be obtained.

Exclusion Criteria:

* systemic disease
* pulp necrosis
* permanent teeth

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children undergoing pulpotomy during regular dental treatment
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Detection of specific inflammatory markers | one year

SECONDARY OUTCOMES:
Pulpotomy failure | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel